CLINICAL TRIAL: NCT01402687
Title: Single Nucleotide Polymorphism (SNP)-Based Prediction of Oral Mucositis Risk in Patients Receiving Hematopoietic Stem Cell Transplants
Brief Title: SNP-Based Prediction of Oral Mucositis Risk in Patients Receiving Hematopoietic Stem Cell Transplants (HSCT)
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Joseph Antin, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 10-236
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Multiple Myeloma
Keywords: Stem Cell Transplant; Mucositis
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Mucositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mucositis Positive: Participants who developed severe mucositis
- Mucositis Negative: Participants who did not develop severe mucositis

SUMMARY:
The goal of this study is to gain new knowledge about genetic risk factors thta may affect the development of mucositis, the chemotherapy-induced sores in the mouth and esophagus following HSCT. The study seeks to understand if different forms of genes result in an increased risk of sores in the mouth and esophagus.

DETAILED DESCRIPTION:
Subjects will be provided with a saliva collection kit which can be used at home. Subjects will return the collection kit in a paid, pre-addressed mailer to the laboratory at Biomodels. The laboratory will isolate and store the DNA located in the cells of the saliva. A portion of this DNA will be used to analyze the different forms of genes. The remainder of the DNA will be destroyed when this study is completed. Biomodels will not be provided with patient identifiers.

The investigators will also collect information from medical records, including information about diagnosis, treatment, stem cell transplantation and post-transplantation outcomes. This information will be de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Have given informed consent to submit a sample of saliva for DNA isolation and SNP analysis
* Have undergone autologous HSCT for treatment of Hodgkin's or non-Hodgkin's lymphoma or multiple myeloma at the Dana-Farber Cancer Institute from 1/1/2006 through 6/30/2010
* Have medical records identifying whether the participants did or did not develop severe mucositis

Exclusion Criteria:

* Received Palifermin (Kepivance) prior to their conditioning regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone autologous HSCT for Hodgkin's or non-Hodgkin's lymphoma or multiple myeloma at Dana Farber Cancer Institute from 1/1/2006 through 6/30/2010.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Develop and validate a clinically applicable SNP-based screening platform for mucositis risk | 2 years
  Develop and validate a clinically applicable SNP-based screening platform that will define mucositis risk among patients undergoing conditioning regimens for HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Antin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States